CLINICAL TRIAL: NCT02269462
Title: Role of Pharmacogenetics in Efavirenz and Nevirapine Pharmacokinetics, Efficacy and Safety in Mother-infant Pairs During Pregnancy and Lactation
Brief Title: A Study to Evaluate the Effects of Genetic Factors on the Pharmacokinetics of Antiretroviral Drugs During Pregnancy and Lactation
Status: Completed | Type: Observational
Sponsor: Adeniyi Olagunju (Other)
Collaborators: University of Liverpool (Other); Obafemi Awolowo University Teaching Hospital (Other)
Responsible Party: Sponsor-Investigator, Adeniyi Olagunju, Lecturer, Obafemi Awolowo University
Organization: Obafemi Awolowo University (Other)
Other Study IDs: BC60000
Record Dates: First submitted 2014-10-02; First posted 2014-10-21 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: HIV; Pregnancy; Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — efavirenz; Nevirapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pregnant women - efavirenz: Pregnant women taking 600 mg efavirenz daily as part of combination antiretroviral therapy for PMTCT and for their own health
  Interventions: Drug: Efavirenz
- Nursing mothers - efavirenz: Nursing mothers taking 600 mg efavirenz daily as part of combination antiretroviral therapy for PMTCT and for their own health and their breastfed babies
  Interventions: Drug: Efavirenz
- Pregnant women - nevirapine: Pregnant women taking 200 mg nevirapine twice daily as part of combination antiretroviral therapy for PMTCT and for their own health
  Interventions: Drug: Nevirapine
- Nursing mothers - nevirapine: Nursing mothers taking 200 mg nevirapine twice daily as part of combination antiretroviral therapy for PMTCT and for their own health and their breastfed babies
  Interventions: Drug: Nevirapine

INTERVENTIONS:
Drug: Efavirenz — 600 mg once daily in combination with other drugs (e.g. tenofovir and emtricitabine)
  Groups: Nursing mothers - efavirenz; Pregnant women - efavirenz
Drug: Nevirapine — 200 mg twice daily in combination with other drugs (e.g. tenofovir and emtricitabine)
  Groups: Nursing mothers - nevirapine; Pregnant women - nevirapine

SUMMARY:
Mother-to-child transmission of HIV (MTCT) during pregnancy and breastfeeding is prevented with maternal antiretroviral drugs (ARV) and infant nevirapine post-exposure prophylaxis (PEP). However, the pharmacokinetics of certain ARVs is associated with marked inter-individual variability. This variability has been associated with single nucleotide polymorphisms (SNPs) in genes encoding metabolising enzymes, transporters and transcriptional regulators. Pregnancy is also associated with additional changes in pharmacokinetics. The resulting sub-therapeutic or supra-therapeutic drug exposures may have serious consequences for virological control, MTCT, emergence of drug resistance, and toxicity. Foetal and infant exposure to maternal ARV during pregnancy and breastfeeding is believed to play a role in the prevention of mother-to-child transmission of HIV (PMTCT). However, such exposures may also result in toxicity. For example, efavirenz is contraindicated in children less than 3 years old or 10kg but transferred to breastfed babies through breast milk. On the other hand, double exposure to nevirapine from breast milk and PEP may also predispose breastfed infants to nevirapine-associated toxicity.

In the proposed study, the influence of selected SNPs in certain drug disposition genes on the pharmacokinetics of efavirenz and nevirapine during pregnancy and lactation, as well as the level of infant exposure to both drugs through breast milk, will be studied. Mathematical models will be developed to predict potential dose optimisation strategies during pregnancy, and to predict infant exposure to maternal drugs through breast milk.

DETAILED DESCRIPTION:
Study design: This is an observational study that will be conducted in two phases. In the preliminary phase, associations between selected SNPs in drug disposition genes and mid-dose plasma and breast milk efavirenz and nevirapine concentrations will be explored in an unselected cohort of HIV positive pregnant women and nursing mothers and their breastfed infants taking either drug as part of combination antiretroviral therapy for PMTCT. In the second phase, the SNP independently associated with the highest predictive power will be used to stratify pregnant women and mother-infant pairs into three groups: non-carriers, heterozygotes, and homozygotes. Randomly selected pregnant women or mother-infant pairs from each group were re-recruited and invited for the intensive pharmacokinetic phase.

Samples collection: In the preliminary phase, mid-dose paired dried blood spots (DBS) (and dried breast milk spots in nursing mothers) samples will be collected at a single, recorded time point post dose. In the intensive pharmacokinetic phase, DBS (and dried breast milk spots in nursing mothers) samples will be collected at multiple time points after an observed dose of efavirenz or nevirapine. Samples will be shipped at room temperature to the Department of Molecular and Clinical Pharmacology, University of Liverpool, United Kingdom for analysis.

DNA extraction and SNP genotyping: Genomic DNA will be extracted using available commercial kits in accordance with the manufacture's protocol and genotyping will be performed by allelic discrimination real-time polymerase chain reaction using TaqMan® chemistry-based assays.

Drug quantification and pharmacokinetic analysis: Liquid chromatography-mass spectrometry methods will be developed for the quantification of efavirenz and nevirapine in DBS and dried breast milk spots. Pharmacokinetic parameters will be determined using standard procedures.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* breastfeeding
* enrolled in PMTCT programme
* started efavirenz- or nevirapine-containing regimen during pregnancy

Exclusion Criteria:

* exclusive replacement feeding
* mixed feeding before 6 months
* severe maternal or infant illness
* maternal or infant treatment with other drugs or herbal medication with known or uncertain interaction with study drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive pregnant women and nursing mothers taking efavirenz or nevirapine as part of HAART to prevent mother-to-child transmission of HIV and/or for their own health and their breastfed infants.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Clearance over systemic availability (Cl/F) during pregnancy. | Patients will be followed for an average of 6 months for the preliminary and intensive pharmacokinetic phase which will occur mainly between the second and third trimester of pregnancy.
Area under the concentration-time curve (AUC0-24 for efavirenz, AUC0-12 for nevirapine) during pregnancy. | Patients will be followed for an average of 6 months for the preliminary and intensive pharmacokinetic phase which will occur mainly between the second and third trimester of pregnancy.
Minimum plasma drug concentration (Cmin) during pregnancy. | Patients will be followed for an average of 6 months for the preliminary and intensive pharmacokinetic phase which will occur mainly between the second and third trimester of pregnancy.
Maximum plasma drug concentration (Cmax) during pregnancy. | Patients will be followed for an average of 6 months for the preliminary and intensive pharmacokinetic phase which will occur mainly between the second and third trimester of pregnancy.
Plasma and breast milk clearance over systemic availability (Cl/F) during lactation. | Pharmacokinetic visits in the preliminary or intensive pharmacokinetic phase will occur mainly from 1 week to 26 weeks postpartum.
Plasma and breast milk area under the concentration-time curve (AUC0-24 for efavirenz, AUC0-12 for nevirapine) during lactation. | Pharmacokinetic visits in the preliminary or intensive pharmacokinetic phase will occur mainly from 1 week to 26 weeks postpartum.
Plasma and breast milk minimum drug concentration (Cmin) during lactation. | Pharmacokinetic visits in the preliminary or intensive pharmacokinetic phase will occur mainly from 1 week to 26 weeks postpartum.
Plasma and breast milk maximum plasma drug concentration (Cmax) during lactation. | Pharmacokinetic visits in the preliminary or intensive pharmacokinetic phase will occur mainly from 1 week to 26 weeks postpartum.

SECONDARY OUTCOMES:
Rate of mother-to-child transmission of HIV. | Infants will be followed up from birth until 18 months of age when all exposure to breastfeeding would have stopped.
Effect of pregnancy on CD4 count change (immunological recovery). | CD4 counts will be determined every 6 months during pregnancy and postpartum, starting from recruitmnent.

CONTACTS AND LOCATIONS:
Overall Officials: Adeniyi Olagunju, Principal Investigator — Obafemi Awolowo University, Nigeria; Andrew Owen, PhD, Principal Investigator — University of Liverpool, United Kingdom
Locations (3):
- Nigeria (3):
  - St Monica's Hospital, Adikpo, Benue State
  - Bishop Murray Medical Centre, Makurdi, Benue State
  - St Mary's Hospital, Okpoga, Benue State

REFERENCES:
- [Result] Olagunju A, Bolaji OO, Amara A, Waitt C, Else L, Soyinka J, Adeagbo B, Adejuyigbe E, Siccardi M, Back D, Owen A, Khoo S. Development, validation and clinical application of a novel method for the quantification of efavirenz in dried breast milk spots using LC-MS/MS. J Antimicrob Chemother. 2015 Feb;70(2):555-61. doi: 10.1093/jac/dku420. Epub 2014 Oct 17. PMID 25326089
- [Result] Olagunju A, Amara A, Waitt C, Else L, Penchala SD, Bolaji O, Soyinka J, Siccardi M, Back D, Owen A, Khoo S. Validation and clinical application of a method to quantify nevirapine in dried blood spots and dried breast-milk spots. J Antimicrob Chemother. 2015 Oct;70(10):2816-22. doi: 10.1093/jac/dkv174. Epub 2015 Jun 24. PMID 26108608
- [Result] Olagunju A, Bolaji O, Amara A, Else L, Okafor O, Adejuyigbe E, Oyigboja J, Back D, Khoo S, Owen A. Pharmacogenetics of pregnancy-induced changes in efavirenz pharmacokinetics. Clin Pharmacol Ther. 2015 Mar;97(3):298-306. doi: 10.1002/cpt.43. Epub 2015 Jan 20. PMID 25669165
- [Result] Olagunju A, Bolaji O, Amara A, Waitt C, Else L, Adejuyigbe E, Siccardi M, Back D, Khoo S, Owen A. Breast milk pharmacokinetics of efavirenz and breastfed infants' exposure in genetically defined subgroups of mother-infant pairs: an observational study. Clin Infect Dis. 2015 Aug 1;61(3):453-63. doi: 10.1093/cid/civ317. Epub 2015 Apr 16. PMID 25882300
- [Result] Olagunju A, Bolaji O, Neary M, Back D, Khoo S, Owen A. Pregnancy affects nevirapine pharmacokinetics: evidence from a CYP2B6 genotype-guided observational study. Pharmacogenet Genomics. 2016 Aug;26(8):381-9. doi: 10.1097/FPC.0000000000000227. PMID 27195527
- [Result] Olagunju A, Khoo S, Owen A. Pharmacogenetics of nevirapine excretion into breast milk and infants' exposure through breast milk versus postexposure prophylaxis. Pharmacogenomics. 2016 Jun;17(8):891-906. doi: 10.2217/pgs-2015-0016. Epub 2016 Jun 7. PMID 27268507
- [Result] Waitt C, Diliiy Penchala S, Olagunju A, Amara A, Else L, Lamorde M, Khoo S. Development, validation and clinical application of a method for the simultaneous quantification of lamivudine, emtricitabine and tenofovir in dried blood and dried breast milk spots using LC-MS/MS. J Chromatogr B Analyt Technol Biomed Life Sci. 2017 Aug 15;1060:300-307. doi: 10.1016/j.jchromb.2017.06.012. Epub 2017 Jun 17. PMID 28651173